CLINICAL TRIAL: NCT04116814
Title: High Resolution Imaging of Retinal Vessels as a Biomarker of Cardiovascular Disease in Patients With Renal Insufficiency - (IRIR)
Brief Title: High Resolution Imaging of Retinal Vessels as a Biomarker of Cardiovascular Disease in Patients With Renal Insufficiency - RI
Acronym: IRIR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Céline FAURE (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-A03143-50
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Retinal Imaging; Cardiovascular Biomarker; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: wall-to-lumen ratio measurement — wall-to-lumen ratio measurement in patients with renal insufficiency

SUMMARY:
The objectives are to better understand, in the dialysis patient, the relationships between microvascular morphometry and cardiovascular events, survival, arterial hypertension, the pathology responsible for renal failure, the age of dialysis and metabolic parameters.

The investigator team also want to better understand the relationship between the diameter of small arteries and parameters such as hypertension, the pathology that causes kidney failure, the age of dialysis, the use of VKA or EPO, metabolic parameters (HbA1c, NFS, reticulocytes, BNP, lipid balance, phosphocalcic balance).

DETAILED DESCRIPTION:
The cardiovascular morbidity of a dialysis patient is 10 times higher than that of a subject in the general population. The patient with renal insufficiency is therefore at high cardiovascular risk. An increase in the wall-to-lumen ratio (WLR) is an early sign of microvascular damage, predictive of the risk of a cardiovascular event. The benefits of WLR measurement are therefore at the level of both the diagnosis and prognosis of vascular disease. Recently, a fundus camera coupled with an adaptive optics system has been able to measure for the first time in vivo non-invasively and reproducibly the wall thickness of the small arteries of the retina, and therefore the WLR, among other biomarkers relating to microvascular remodelling.

Studies in hypertension have confirmed that the rtX1 camera allows reliable and reproducible measurements of the WLR. The main aim of our study is to evaluate the value of the WLR as a biomarker of the risk of cardiovascular morbidity and mortality in patients with renal insufficiency.

The objectives are to better understand, in the dialysis patient, the relationships between microvascular morphometry and cardiovascular events, survival, arterial hypertension, the pathology responsible for renal failure, the age of dialysis and metabolic parameters.

The investigator team also want to better understand the relationship between the diameter of small arteries and parameters such as hypertension, the pathology that causes kidney failure, the age of dialysis, the use of VKA or EPO, metabolic parameters (HbA1c, NFS, reticulocytes, BNP, lipid balance, phosphocalcic balance).

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patients with renal insufficiency: waiting for management (dialysis or transplant), during dialysis or after a kidney transplant followed in the nephrology department of the Saint Martin clinic.
* First examination in adaptive optics giving a usable result (possibility of measuring the WLR)
* Affiliate or beneficiary of a social security scheme
* Patient having given their free and informed consent

Exclusion Criteria:

* Protected patients: adults under guardianship, trusteeship or other legal protection, deprived of liberty by judicial or administrative decision, hospitalised without consent.
* Pregnant, lactating or parturient women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient included with Ophthalmological examination with WLR measurement in adaptive optics
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2022-03-29 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Predictibilty of WLR | 3 years
  The primary endpoint is time to event (cardiovascular events or death) in months, assessed by survival analysis.

SECONDARY OUTCOMES:
WLR associated biomarker | 3 years
  Secondary endpoints:
  - Association between WLR and cardiovascular risk factors, medical history and metabolic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Martin Private Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided